CLINICAL TRIAL: NCT04418830
Title: A Prospective, Multicenter Study Evaluating the Safety and Performance of Interbody Implants for the Treatment of Patients With Degenerative Conditions of the Thoracic and/or Lumbar Spine
Brief Title: Lumbar Interbody Implant Study
Status: Enrolling by invitation | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.LIB1119
Record Dates: First submitted 2020-06-02; First posted 2020-06-05 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Degenerative Disc Disease; Degenerative Spondylolisthesis; Degenerative Scoliosis; Spinal Stenosis; Sagittal Deformity
Keywords: Spine Surgery; Medical Device
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: US Export: Yes

GROUPS / COHORTS (14):
- Base Interfixated System
- Brigade Interfixated System
- Coalesce Thoracolumbar Interbody
- Cohere XLIF Interbody System
- CoRoent Ti PLIF Interbody System
- CoRoent Ti TLIF Interbody System
- MLX - Medial Lateral Expandable Interbody System
- Modulus TLIF Interbody System
- Modulus XLIF Interbody System
- TLX Interbody System
- XLX ACR Interbody System
- CoRoent Ti XLIF Interbody System
- Cohere TLIF
- Modulus ALIF

SUMMARY:
The objective of this study is to evaluate the safety and performance of NuVasive interbody implants when used during thoracic and/or lumbar spine surgery as measured by reported complications, radiographic outcomes, and patient-reported outcomes. This study is being undertaken to identify possible residual risks and to clarify mid- to long-term clinical performance that may affect the benefit/risk ratios of these interbody implants.

DETAILED DESCRIPTION:
This study is a prospective, uncontrolled, multicenter study to evaluate the safety and performance of select interbody implant devices in patients who undergo interbody fusion surgery. Consecutive patients at a given site who meet eligibility requirements will be asked to consent to participate in the study. These patients will present with degenerative conditions in the thoracic and/or lumbar spine that are amenable to surgical treatment and will be screened prior to study enrollment. Once enrolled into the study, subjects will undergo interbody fusion surgery using one of the NuVasive interbody implant groups based on the surgeon's standard of care. At least 1050 subjects (a minimum of 75 patients in each implant group) will be enrolled and will be followed for 24 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are ≥18 years of age at the time of consent
2. Planned spine surgery using interbody implants at:

   1. One or two adjacent thoracic, lumbar, and/or lumbosacral levels for degenerative disc disease or degenerative spondylolisthesis, or
   2. One or two adjacent thoracic, lumbar, and/or lumbosacral levels for spinal stenosis (not applicable for MLX, TLX, or XLX ACR), or
   3. Any number of thoracic, lumbar, and/or lumbosacral levels for degenerative scoliosis (defined as >10º coronal curve), or
   4. Any number of thoracic, lumbar, and/or lumbosacral levels for sagittal deformity (not applicable for MLX, TLX, or XLX ACR).
3. Use of one of the following implants (NuVasive, Inc., San Diego, CA):

   1. Base Interfixated
   2. Brigade Interfixated
   3. Coalesce Thoracolumbar
   4. Cohere TLIF
   5. Cohere XLIF
   6. Coroent Ti PLIF
   7. Coroent Ti TLIF
   8. Coroent Ti XLIF
   9. MLX
   10. Modulus ALIF
   11. Modulus TLIF
   12. Modulus XLIF
   13. TLX
   14. XLX ACR
4. Interbody fusion with one or more of the following (as allowed by implant type):

   1. autograft
   2. allograft (i.e., cancellous and/or corticocancellous allograft bone)
   3. Attrax Putty (NuVasive) (not applicable for MLX, TLX, or XLX ACR)
5. NuVasive supplemental internal fixation cleared by the applicable regulatory body for use in the thoracolumbar spine (unless the interbody device to be used is interfixated and is cleared by the regulatory body to be used standalone)
6. Able to undergo surgery based on physical exam, medical history, and surgeon judgment
7. Understands the conditions of enrollment, is willing to follow medical advice including postoperative activity restrictions per the surgeon's standard of care, and is willing to sign an informed consent form to participate in the study

Exclusion Criteria:

1. Use of any bone graft that is not cleared by the applicable regulatory body for use within interbody implants. Examples of these include:

   1. Bone morphogenetic protein (BMP) (e.g., Infuse (Medtronic))
   2. Synthetic bone graft extenders (e.g., Attrax Scaffold (NuVasive), Formagraft (NuVasive), Mastergraft (Medtronic), Vitoss (Stryker), Actifuse (Baxter), nanOss (RTI Surgical), Fibergraft (Prosidyan/Depuy Synthes), ChronOs (Depuy Synthes))
   3. Demineralized bone matrices (DBM) regulated as medical devices by the FDA (e.g., Grafton Putty/Gel (Medtronic), DBX (MTF/Depuy Synthes), Accell Evo3 (IsoTis), Propel Putty/Gel (NuVasive))
   4. Peptide enhanced bone graft (e.g., iFactor (Cerapedics))
2. Previous lumbar fusion surgery at the level(s) to be treated (adjacent level surgery is acceptable; prior decompression is acceptable)
3. Patient is involved in active litigation relating to the spine (worker's compensation claim is allowed if it is not contested)
4. Use of bone growth stimulators postoperatively
5. Active smoking within 6 weeks before surgery
6. Patient has known sensitivity to the materials implanted
7. Systemic or local infection (latent or active) or signs of local inflammation
8. Patient has inadequate bone stock or bone quality, or a physical or medical condition that would prohibit beneficial surgical outcomes based on surgeon judgment
9. Patient is a prisoner
10. Patient is participating in another clinical study that would confound study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Enrolled Population will include all subjects who meet the criteria for enrollment, specifically, those subjects who:
  * Satisfied the inclusion and exclusion criteria
  * Signed the informed consent
  * Underwent the surgical procedure, as defined in this protocol
  Subjects not meeting any of these criteria will not be considered enrolled in the study, and therefore not included in any study population or analysis.
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Complications of Interbody Implants | 24 months
  Rate of complications attributable to the use of the interbody implants to be studied
Radiographic Fusion Success | 24 months
  The proportion of subjects with apparent radiographic fusion at or before 24 months within each treatment group

SECONDARY OUTCOMES:
Percentage of subjects meeting minimal clinically important difference (MCID) as compared to baseline for back/leg pain measured by visual analog scale (VAS). | 24 months
  Back and leg pain measured using a visual analog scale (VAS) will be assessed to determine the percentage of subjects who meet MCID (1.2 points and 1.6 points respectively) where 0 is "No Pain" and 10 is "Unbearable Pain".
Percentage of subjects meeting minimal clinically important difference (MCID) as compared to baseline for disability measured by the Oswestry disability index. | 24 months
  Disability measured by the Oswestry disability index (ODI) will be assessed to determine the percentage of subjects who meet MCID (12.8 points) where a higher score on the ODI indicates a more severe disability.
Percentage of subjects meeting minimal clinically important difference (MCID) as compared to baseline measured by overall physical and mental health from PROMIS-10. | 24 months
  Overall physical and mental health measured by PROMIS-10 will be assessed to determine the percentage of subjects who meet MCID (5 points). PROMIS-10 scoring uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
Complications attributable to the use of any additional NuVasive instruments, implants, or technologies | 24 months
  Rate of complications attributable to the use of any additional NuVasive instruments, implants, or technologies

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Malone, MS, Study Director — Globus Medical
Locations (16):
- United States (16):
  - University of California San Diego, La Jolla, California
  - Verma Spine, Los Alamitos, California
  - Valley Spine Care, Merced, California
  - Hoag Orthopedics, Orange, California
  - Hartford Healthcare Bone and Joint Institute, Hartford, Connecticut
  - Lyerly Neurosurgery, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - DuPage Medical Group, Naperville, Illinois
  - Beaumont Hospital Research Institute, Royal Oak, Michigan
  - Columbia Orthopaedics Group, Columbia, Missouri
  - Duke University, Durham, North Carolina
  - Atlantic Brain and Spine, Wilmington, North Carolina
  - Summa Health, Akron, Ohio
  - Ohio State University, Dublin, Ohio
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No